CLINICAL TRIAL: NCT01973010
Title: Phase 1 Study of Massage Therapy for Chronic Low Back Pain
Brief Title: Massage Therapy for Chronic Low Back Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011SZ0302.1
Record Dates: First submitted 2013-10-22; First posted 2013-10-31 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Low Back Pain
Keywords: massage; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Massage; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Massage (Experimental): To treat low back pain with massage
  Interventions: Other: Massage
- Ibuprofen (Active Comparator): Medicine control group
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Other: Massage — Massage therapy is an intervention that can be used to relax muscle and regulate displaced joints by manual manipulation.
  Other Names: Tuina
  Arms: Massage
Drug: Ibuprofen — Ibuprofen is an common analgesics which has been widely used in regular control of various pain symptom.
  Other Names: Pain killer
  Arms: Ibuprofen

SUMMARY:
The purpose of this study is to determine whether massage is effective in the treatment of low back pain and to optimize clinical therapeutic schedule of massage for low back pain.

DETAILED DESCRIPTION:
Chronic low back pain is a prevalent condition among adults. Large majority of the population suffer from Chronic low back pain in their lifetime. At present, there is still no standard treatment for chronic low back pain. Massage is commonly chose and widely used by sufferer as a complement to conventional treatment. However, its effectiveness is still not convinced. This trial is designed to assess the effectiveness of massage for chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* In accordance of the diagnostic criteria of low back pain;
* Age between 20 and 55 years old;
* Not taking hormone drugs or antirheumatic drugs within the latest 2 months;
* No allergy history of hormone drugs Pain medicine;
* volunteer participation and signing an informed consent in writing.

Exclusion Criteria:

* Being pregnant or during lactation;
* Having suffered from serious psychiatric, neurologic, cardiovascular, respiratory, or renal illnesses, and so forth;
* Severe neurological deficits caused by severe lumbar disc protrusion, and operation indications;
* Receiving message therapy in past 3 months for releasing low back pain.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Back function measured by Roland-Morris Disability Questionnaire at 2 months | At baseline, 4th, 6th, 8th week
  to assess the recovery of back function

SECONDARY OUTCOMES:
Japanese Orthopaedic Association Scores | At baseline, 4th, 6th, 8th week
  to assess the improvement of back function
McGill pain questionnaire | At baseline, 4th, 6th, 8th week
  To assess the alleviation of pain

CONTACTS AND LOCATIONS:
Overall Officials: Fanrong Liang, Professor, Principal Investigator — Chengdu University of TCM
Locations (1):
- Acupuncture and Tuina college of Chengdu University of TCM, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Yang M, Feng Y, Pei H, Deng S, Wang M, Xiao X, Zheng H, Lai Z, Chen J, Li X, He X, Liang F. Effectiveness of Chinese massage therapy (Tui Na) for chronic low back pain: study protocol for a randomized controlled trial. Trials. 2014 Oct 29;15:418. doi: 10.1186/1745-6215-15-418. PMID 25352050